CLINICAL TRIAL: NCT03648190
Title: Evaluation of Platelet Surface Glycoproteins in Patients With Inherited Thrombocytopathy: Association With Aggregation Studies and Bleeding Severity
Brief Title: Platelet Glycoproteins in Inherited Thrombocytopathy: Association With Aggregation Studies and Bleeding Severity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Ashraf, Assistant Lecturer, Assiut University
Other Study IDs: 17200237
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Bleeding; Platelet Dysfunction
Keywords: GT; CD
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inherited qualitative platelets defect: Clinical manifestations in the form of mucocutaneous bleeding or hemorrhage.
  Bleeding patients with acquired bleeding disorders, coagulation defects, and those on antiplatelet drugs will be excluded from the study.
  Interventions: Diagnostic Test: Flowcytometry analysis of platelets surface receptors
- Control: Normal healthy participants, with no manifestations of bleeding disorders.
  Interventions: Diagnostic Test: Flowcytometry analysis of platelets surface receptors

INTERVENTIONS:
Diagnostic Test: Flowcytometry analysis of platelets surface receptors — BD FACSCalibur flowcytometry instrument.
  Platelet flow cytometry is an emerging tool in diagnostic and therapeutic hematology. It is eminently suited to study the expression of platelet surface receptors both qualitatively as well as quantitatively.
  Flow cytometry rapidly measures the specific characteristics of a large number of cells in suspension. Typically, the cells are labeled with fluorescently conjugated monoclonal antibodies (mAbs).
  Other Names: Platelets aggregation tests by aggregometer

SUMMARY:
Disorders of platelet function are characterized by variable mucocutaneous bleeding manifestations and excessive hemorrhage following surgical procedures or trauma. Generally, most patients have mild to moderate bleeding manifestations with a prolonged bleeding time.

Platelet aggregation and secretion studies using platelet-rich plasma (PRP) provide evidence for platelet dysfunction but are neither predictive of severity of clinical manifestations nor the molecular mechanisms.

Glanzmann's thrombasthenia (GT) is a rare autosomal recessive genetic bleeding syndrome characterized by defects in platelet aggregometry. The clinical phenotype of patients with GT is variable. Some suffer from severe bleeding, while others have only mild bleeding. Some studies found bleeding severity in GT was influenced by the abundance and functioning of platelet receptors involved in aggregation and adhesion.

In addition to a complete medical history, a GT diagnosis requires a comprehensive laboratory workup, including platelet aggregation analysis, and a confirmation by flowcytometry or western blotting with monoclonal antibodies that recognize the GPIIb/IIIa complex.

Platelet flow cytometry is an emerging tool in diagnostic and therapeutic hematology. It is eminently suited to study the expression of platelet surface receptors both qualitatively as well as quantitatively.

Aim of the study:-

* Determine the role of flowcytometry as a quantitative measurement tool of platelets surface glycoproteins in patients with inherited thrombocytopathies and its correlation with bleeding severity of these patients.
* To compare the efficacy, advantages and disadvantages between platelets flowcytometry and aggregometer in diagnosing various inherited thrombocytopathies.

DETAILED DESCRIPTION:
This study is a case-control observational study to be done at Clinical pathology department, Assiut University hospital, Assiut University, Egypt.

Patients with inherited qualitative platelets defect with clinical manifestations in the form of mucocutaneous bleeding or hemorrhage will be included in the study. Individuals with similar age and sex distribution to the patient group will act as controls. Control group shouldn't take medications or anti-platelet drugs for the preceding two weeks. They should have normal platelet count and morphology. Bleeding patients with acquired bleeding, coagulation defects, and those on anti-platelet drugs will be excluded from the study.

All Patients with inherited platelets function disorders will be subjected to:-

I - Careful history and clinical examination data collecting including:

Clinical history of bleeding such as (Sites, Severity and frequency of bleeding, trauma related events, history of surgical procedures, history of menorrhagia in females, history of packed red cell/ platelets transfusion.

II - Family history such as consanguinity, bleeding complications in any parents/ siblings.

III - Grading of bleeding severity: according to World Health Organization (WHO) bleeding assessment scale from grade 1 to grade 4.

The following routine investigations will be done:-

1. Complete blood count (CBC) analysis.
2. Prothrombin time, concentration and international normalized ratio (INR) assay.
3. Activated partial thromboplastin time assay.
4. Fibrinogen level and thrombin time assay.

The following specific investigations:-

1. Platelets aggregation tests by aggregometer using four different agonists (ADP, Collagen, Arachidonic acid and ristocetin) on Bio/Data PAP-8E.
2. Flowcytometry analysis of platelets receptors (CD 41, CD 61 and CD 42b) on BD FACSCalibur flowcytometry instrument.

Data collection and analysis will be done by computer program SPSS version 21 Chicago USA. Data expressed as mean ±SD, mean±SE, number and percentage. Using Manwhitny test to determine the significance for numeric variable and chisquare to determine the significance for non-parametric variable. ROC curve was done to determine the area under curve (AUC), sensitivity and specificity for each marker.

ELIGIBILITY:
Inclusion Criteria:

* Bleeding patients.

Exclusion Criteria:

* Coagulation defects, and those on anti-platelet drugs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Bleeding patients suffering from inherited qualitative platelets defect, with the exclusion of coagulation defects, acquired bleeding disorders and anti-platelet drugs intake. Both male and females are eligible with no age limits.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Establishment of a protocol for Flowcytometry device to be used in routinely diagnosing cases with inherited platelets function defects. | 6 Weeks
  Determine the ability of flowcytometry to assay (determine the levels of expression of each surface marker in percent) platelets surface glycoproteins (CD 41, CD 61 and CD 42b) using BD FACSCalibur flowcytometry instrument in patients with inherited thrombocytopathies and its correlation with bleeding severity of these patients with establishment of a protocol for it to be used in routinely diagnosing these cases.

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Galal, MD, Principal Investigator — Assiut University; Madleen Adel, MD, Study Chair — Assiut University; Eman Nasr-Eldin, MD, Study Chair — Assiut University; Mohammed Ashraf, M.Sc, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou L, Jiang M, Shen H, You T, Ding Z, Cui Q, Ma Z, Yang F, Xie Z, Shi H, Su J, Cao L, Lin J, Yin J, Dai L, Wang H, Wang Z, Yu Z, Ruan C, Xia L. Clinical and molecular insights into Glanzmann's thrombasthenia in China. Clin Genet. 2018 Aug;94(2):213-220. doi: 10.1111/cge.13366. Epub 2018 May 22. PMID 29675921
- [Background] Harrison P. Assessment of platelet function in the laboratory. Hamostaseologie. 2009 Jan;29(1):25-31. PMID 19151842
- [Background] Saboor M, Moinuddin M, Ilyas S. New horizons in platelets flow cytometry. Malays J Med Sci. 2013 Mar;20(2):62-6. PMID 23983579